CLINICAL TRIAL: NCT00825747
Title: Clinical Evaluation of the Aspheric SeeLens AF Intra-ocular Lens.
Brief Title: Evaluation of Seelens AF, an Aspheric Intra-ocular Lens
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study was closed
Sponsor: Hanita Lenses (Industry)
Responsible Party: Simha Siboni, regulatory manager, Hanita Lenses, Israel
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SeeLensAF 65
Record Dates: First submitted 2009-01-18; First posted 2009-01-21 (Estimated); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Cataract
Keywords: Cataract; Cataract surgery; intraocular lens; Aspheric lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: SeeLens AF intra-ocular lens — the SeeLens AF is an acrylic hydrophilic C shaped haptics intra-ocular lens, designed for implantation in the lenticular capsular bag or the sulcus during cataract surgery.
  Other Names: aspheric SeeLens

SUMMARY:
Senile cataract is managed by cataract extraction and intra-ocular lens (IOL) implantation. The purpose of this study is to evaluate the safety and efficacy of the SeeLens AF, an acrylic hydrophilic aspheric IOL. This lens was designed to reduce vision aberrations and secondary cataract formation rate.

Preoperative evaluation: Best corrected visual acuity, refraction, comprehensive slit lamp examination and biometry.

Surgical procedure: Cataract surgery using a clear corneal incision (1.8mm to2.4mm), phacoemulsification and implantation of the SeeLens AF to the capsular bag. IOL implantation parameters will be evaluated by the surgeon.

Postoperative follow up: Best corrected visual acuity, uncorrected visual acuity, refraction and comprehensive slit lamp examinations up to 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Senile Cataract
* Age >18 years
* Cataract extraction using phacoemulsification
* Corneal incision less than 1.5 mm

Exclusion Criteria:

* Allergy/sensitivity to eye drops used during and after cataract surgery
* Amblyopia/ strabismus
* Ocular disease, other than cataract, diminishing visual acuity, such as corneal opacity, advanced glaucoma, diabetic retinopathy, exudative or moderate to severe non-exudative age-related macular degeneration, uveitis.
* previous ocular surgery or ocular trauma in the investigated eye
* Ocular anomaly, such as microphthalmos
* Keratometry values less than 40 diopters or more than 47 diopters.
* Ocular axial length less than 21.0 mm or longer than 25.0 mm
* Intra-operative complications prior to intraocular lens implantation, such as tear of the posterior capsule.
* posterior capsular scar
* visual acuity in the fellow eye less than 20/200

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity 3 months after SeeLens AF implantation | 3 months

SECONDARY OUTCOMES:
Complications related to SeeLens AF implantation during cataract surgery. | 3 months
Postoperative severe intra-ocular inflammation or infection | 3 months
Prediction of ocular refraction after cataract surgery with Seelens AF implantation | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yokrat Ton, MD, Principal Investigator — Meir Medical Center, affiliated with Tel-Aviv University, Tel-Aviv, Israel
Locations (2):
- Israel (2):
  - Soroka University Medical Center, Beersheba
  - Meir Medical Center, Kfar Saba